CLINICAL TRIAL: NCT03258762
Title: A Single Centre, Open-label, Parallel-group, Single Oral Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Pyrimethamine in Healthy Japanese and Caucasian Male Subjects
Brief Title: Phase I Study of Pyrimethamine in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204678
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2019-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Toxoplasmosis
Keywords: Japanese; Caucasian; pharmacokinetics; pyrimethamine; toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis | interventions — Pyrimethamine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Japanese male subjects (Experimental): Healthy Japanese male subjects will receive a single oral dose of Pyrimethamine 50 mg in the fasted state co-administered with calcium folinate 15 mg on Day 1. Oral calcium folinate will be administered once daily until Day 8. Blood samples for PK analysis will be collected prior to administering first dose of Pyrimethamine and over 22 days post dose. Each subject will participate in the study for a duration of approximately 2 months from screening to follow-up.
  Interventions: Drug: Pyrimethamine; Drug: Calcium folinate
- Healthy Caucasian male subjects (Experimental): Healthy Caucasian male subjects will receive a single oral dose of Pyrimethamine 50 mg in the fasted state co-administered with calcium folinate 15 mg on Day 1. Oral calcium folinate will be administered once daily until Day 8. Blood samples for PK analysis will be collected prior to administering first dose of Pyrimethamine and over 22 days post dose. Each subject will participate in the study for a duration of approximately 2 months from screening to follow-up.
  Interventions: Drug: Pyrimethamine; Drug: Calcium folinate

INTERVENTIONS:
Drug: Pyrimethamine — Pyrimethamine will be available as 25 mg tablets. Subjects will be orally administered two pyrimethamine tablets on Day 1 in a fasted condition with 240 mL of water.
Drug: Calcium folinate — Calcium folinate will be available as 5 mg tablets. Subjects will be orally administered three calcium folinate tablets on Day 1 along with pyrimethamine followed by once daily administration of calcium folinate until Day 8. Each administration will be with 240 mL water.

SUMMARY:
Pyrimethamine in combination with a sulphonamide is known to be effective in the treatment of toxoplasmosis. However, Pyrimethamine has not been approved by the Japanese regulatory body (Pharmaceutical and Medical Devices Agency [PMDA]/ Ministry of Health, Labor and Welfare [MHLW]). The pharmacokinetics (PK) of Pyrimethamine has been investigated following administration of Sulfadoxine/Pyrimethamine tablet in healthy Japanese subjects. However, the study did not provide sufficient information for approval of Pyrimethamine in Japan; hence, PMDA has requested confirmation of the PK of Pyrimethamine in another PK study in Japanese and Caucasian healthy subjects. This study will be a single centre, open-label, parallel-group, single oral dose study to evaluate the PK, safety and tolerability of Pyrimethamine in healthy Japanese and Caucasian male subjects. Subjects will undergo a screening visit within 30 days prior to first dose of the study drug. On Day 1, subjects will be administered a single oral dose of pyrimethamine 50 milligrams (mg) along with calcium folinate 15 mg after an overnight fast of at least 10 hours. Subjects will continue to receive calcium folinate once daily until Day 8 of the treatment period. Blood sampling for PK analysis and safety assessments will be performed prior to dosing and over 22 days after dosing. Each subject will participate in the study for approximately 2 months from screening to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be between 20 and 64 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 18.5 to 30.0 kilogram per square meters (kg/m^2) (inclusive).
* Japanese or Caucasian male.
* A male subject must agree to use contraception during the treatment period and until follow-up.
* Japanese ethnic origin defined as having been born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Subjects should also have lived outside Japan for less than 10 years at the time of screening.
* Caucasian subject will be defined as an individual having four grandparents who are all descendants of the original people of Europe.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions of the study.

Exclusion Criteria:

* Alanine aminotransferase (ALT) > 1.5 times upper limit of normal (ULN).
* Bilirubin > 1.5 times ULN (isolated bilirubin > 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35 percent).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 milliseconds (msec).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* Hematological values: outside normal range at screening.
* Serum creatinine level: outside normal range at screening visit.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days before signing of consent in this clinical study involving an investigational study treatment or any other type of medical research.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment. Test is optional and subjects with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as: For an average weekly intake of > 14 units for males. One unit is equivalent to 10 grams (g) of alcohol: a can of mid-strength (equivalent to 375 mL) beer, 1 glass (100 mL) of table wine or 1 measure (30 mL) of spirits (including rice wine).
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-11-19 (Actual); Study Completion 2017-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20305

REFERENCES:
- [Background] Iida T, Nand RA, Ino H, Ogura H, Itoh H, Igarashi H, Numachi Y, Gross AS. Evaluation of the Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of Pyrimethamine in Healthy Male Subjects of Japanese and European Ancestry. Clin Pharmacol Drug Dev. 2020 Aug;9(6):768-773. doi: 10.1002/cpdd.771. Epub 2020 Jan 16. PMID 31950646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in healthy Japanese and Caucasian male participants to evaluate safety, tolerability and pharmacokinetic (PK) parameters of Pyrimethamine. This study was conducted at a single center in Australia.
Pre-assignment Details: A total of 14 healthy participants were enrolled in this study.
Groups:
- Healthy Japanese Participants: Healthy Japanese male participants received a single oral dose of Pyrimethamine 50 milligram (mg) tablet in the fasted state co-administered with calcium folinate 15 mg tablet on Day 1. Oral calcium folinate was administered once daily until Day 8 along with 240 milliliters (mL) of water.
- Healthy Caucasian Participants: Healthy Caucasian male participants received a single oral dose of Pyrimethamine 50 mg tablet in the fasted state co-administered with calcium folinate 15 mg tablet on Day 1. Oral calcium folinate was administered once daily until Day 8 along with 240 mL of water.
Period: Overall Study
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Japanese Participants: Healthy Japanese male participants received a single oral dose of Pyrimethamine 50 mg tablet in the fasted state co-administered with calcium folinate 15 mg tablet on Day 1. Oral calcium folinate was administered once daily until Day 8 along with 240 mL of water.
- Total: Total of all reporting groups
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (3.27) | 30.7 (6.02) | 29.9 (4.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian: Japanese Heritage/East Asian | 7 | 0 | 7
  White/Caucasian/European heritage | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis. PK Population is defined as all participants who administered at least one dose of study treatment and who have PK sample taken and analyzed.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Nanogram per milliliter | 430.5 (13.3)

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC[0-t]) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 59013.1 (15.3)

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 64670.3 (16.6)

4. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 (AUC[0-24]) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 8756.3 (8.0)

5. Primary Outcome: Terminal Half-life (t1/2) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Hours | 122.75 (21.499)

6. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Hours | 2.000 [1.00 to 6.00]

7. Primary Outcome: Apparent Clearance Following Oral Dosing (CL/F) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Milliliter per hour | 773.2 (16.6)

8. Primary Outcome: Apparent Volume of Distribution Following Oral Dosing (Vd/F) of Pyrimethamine in Healthy Japanese Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter
Arm/Group | Healthy Japanese Participants
Number analyzed (Participants) | 7
Milliliter | 135330.9 (5.5)

9. Secondary Outcome: Cmax of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Nanogram per milliliter | 371.1 (10.0)

10. Secondary Outcome: AUC (0-t) of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 41582.0 (26.9)

11. Secondary Outcome: AUC (0-inf) of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 44869.1 (27.0)

12. Secondary Outcome: AUC (0-24) of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Hours* nanogram per milliliter | 6930.8 (19.3)

13. Secondary Outcome: Tmax of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Hours | 1.000 [1.000 to 6.00]

14. Secondary Outcome: T1/2 of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Hours | 99.46 (20.745)

15. Secondary Outcome: CL/F of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per hour
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Milliliters per hour | 1114.4 (27.0)

16. Secondary Outcome: Vd/F of Pyrimethamine in Healthy Caucasian Male Participants
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 6, 12 hours post-dose on Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters
Arm/Group | Healthy Caucasian Participants
Number analyzed (Participants) | 7
Milliliters | 157125.8 (16.8)

17. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or events associated with liver injury and impaired liver function were categorized as SAE. All participants who take at least one dose of study treatment were included in Safety Population.
Time Frame: Up to Day 23
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Participants
  Any AEs | 2 | 6
  Any SAEs | 0 | 0

18. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters: Glucose, Sodium, Calcium, Potassium, and Urea.
Description: Blood samples were collected for the analysis of clinical chemistry parameters including glucose, sodium, calcium, potassium, and urea at indicated time points. Day -1 value was defined as Baseline for clinical chemistry parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Millimoles per liter
  Glucose, 24 hours, n=7, 7 | -0.33 (0.403) | -0.26 (0.310)
  Glucose, 96 hours, n=7, 7 | -0.43 (0.281) | -0.10 (0.200)
  Glucose, 168 hours, n=7, 7 | -0.60 (0.424) | -0.37 (0.214)
  Category title 4. : Glucose, 336 hours, n=7, 7 | -0.43 (0.335) | -0.09 (0.241)
  Glucose, Follow-up (504 hours), n= 7, 6: number analyzed (Participants) | 7 | 6
  Glucose, Follow-up (504 hours), n= 7, 6 | -0.24 (0.395) | 0.00 (0.276)
  Calcium, 24 hours, n=7, 7 | -0.116 (0.0608) | -0.054 (0.0862)
  Calcium, 96 hours, n=7, 7 | -0.006 (0.0947) | -0.033 (0.0670)
  Calcium, 168 hours, n=7, 7 | -0.006 (0.0730) | -0.033 (0.0739)
  Calcium, 336 hours, n=7, 7 | -0.083 (0.1224) | -0.040 (0.0432)
  Calcium, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Calcium, Follow up (504 hours), n=7, 6 | -0.100 (0.0781) | -0.042 (0.0637)
  Potassium, 24 hours, n=7, 7 | -0.03 (0.427) | 0.00 (0.580)
  Potassium, 96 hours, n=7, 7 | 0.00 (0.356) | -0.11 (0.515)
  Potassium, 168 hours, n=7, 7 | 0.01 (0.463) | -0.21 (0.241)
  Potassium, 336 hours, n=7, 7 | -0.10 (0.216) | -0.21 (0.515)
  Potassium, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Potassium, Follow up (504 hours), n=7, 6 | 0.09 (0.402) | -0.22 (0.488)
  Sodium, 24 hours, n=7, 7 | -0.3 (3.55) | 0.0 (2.83)
  Sodium, 96 hours, n=7, 7 | -0.6 (3.05) | 1.0 (1.73)
  Sodium, 168 hours, n=7, 7 | -1.3 (2.63) | 1.7 (1.25)
  Sodium, 336 hours, n=7, 7 | 0.3 (1.38) | -0.3 (1.38)
  Sodium, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Sodium, Follow up (504 hours), n=7, 6 | -0.1 (1.86) | -0.5 (1.76)
  Urea, 24 hours, n=7, 7 | 0.33 (0.772) | 1.01 (1.110)
  Urea, 96 hours, n=7, 7 | 0.26 (1.190) | -0.03 (0.660)
  Urea, 168 hours, n=7, 7 | 0.41 (1.053) | -0.26 (0.885)
  Urea, 336 hours, n=7, 7 | -0.16 (0.896) | 1.06 (1.726)
  Urea, Follow up,(504 hours) n=7, 6: number analyzed (Participants) | 7 | 6
  Urea, Follow up,(504 hours) n=7, 6 | 0.99 (1.995) | 1.27 (1.317)

19. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters: Alkaline Phosphatase, Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including alkaline phosphatase, ALT and AST at indicated time points. Day -1 value was defined as Baseline for clinical chemistry parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
International units per liter
  Alkaline Phosphatase, 24 hours, n=7, 7 | -9.0 (11.60) | -3.3 (5.71)
  Alkaline Phosphatase, 96 hours, n=7, 7 | -6.7 (10.67) | -3.1 (2.97)
  Alkaline Phosphatase, 168 hours, n=7, 7 | -7.0 (11.56) | -4.1 (3.48)
  Alkaline Phosphatase, 336 hours, n=7, 7 | -11.0 (12.00) | -2.9 (5.90)
  Alkaline Phosphatase, Follow-up (504 hours), n=7,6: number analyzed (Participants) | 7 | 6
  Alkaline Phosphatase, Follow-up (504 hours), n=7,6 | -9.6 (11.18) | -9.3 (5.89)
  ALT, 24 hours, n=7, 7 | -3.0 (5.03) | -3.3 (2.81)
  ALT, 96 hours, n=7, 7 | -2.1 (6.23) | -5.1 (4.91)
  ALT, 168 hours, n=7, 7 | 0.7 (5.53) | -4.4 (8.16)
  ALT, 336 hours, n=7, 7 | 0.9 (9.84) | -3.9 (2.79)
  ALT, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  ALT, Follow up (504 hours), n=7, 6 | 0.4 (11.25) | -5.3 (4.59)
  AST, 24 hours, n=7, 7 | -3.4 (4.61) | -1.9 (4.56)
  AST, 96 hours, n=7, 7 | -3.7 (5.12) | -4.3 (6.55)
  AST, 168 hours, n=7, 7 | -2.0 (5.32) | -3.0 (7.62)
  AST, 336 hours, n=7, 7 | 0.3 (9.81) | -2.4 (5.86)
  AST, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  AST, Follow up (504 hours), n=7, 6 | 0.0 (4.16) | -1.5 (6.83)

20. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters: Direct Bilirubin, Bilirubin, Creatinine.
Description: Blood samples were collected for the analysis of clinical chemistry parameters including direct bilirubin, bilirubin and creatinine at indicated time points. Day -1 value was defined as Baseline for clinical chemistry parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Micromoles per liter
  Direct bilirubin, 24 hours, n=7, 7 | 0.7 (1.98) | 0.6 (0.53)
  Direct bilirubin, 96 hours, n=7, 7 | 0.4 (1.27) | 0.7 (1.70)
  Direct bilirubin, 168 hours, n=7, 7 | 0.6 (2.30) | 0.9 (1.35)
  Direct bilirubin, 336 hours, n=7, 7 | -0.3 (1.60) | 0.9 (1.95)
  Direct bilirubin, Follow-up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Direct bilirubin, Follow-up (504 hours), n=7, 6 | -0.3 (1.50) | 0.3 (1.97)
  Bilirubin, 24 hours, n=7, 7 | 1.4 (5.16) | 3.1 (4.56)
  Bilirubin, 96 hours, n=7, 7 | -0.6 (5.83) | 2.4 (5.47)
  Bilirubin, 168 hours, n=7, 7 | 0.7 (8.10) | 1.0 (5.23)
  Bilirubin, 336 hours, n=7, 7 | -4.0 (5.83) | -0.3 (5.22)
  Bilirubin, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Bilirubin, Follow up (504 hours), n=7, 6 | -3.4 (5.56) | -1.7 (7.06)
  Creatinine, 24 hours, n=7, 7 | 21.7 (8.16) | 26.6 (6.68)
  Creatinine, 96 hours, n=7, 7 | 24.4 (5.06) | 30.1 (7.84)
  Creatinine, 168 hours, n=7, 7 | 20.9 (5.08) | 24.6 (4.83)
  Creatinine, 336 hours, n=7, 7 | 14.1 (6.18) | 14.9 (4.71)
  Creatinine, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Creatinine, Follow up (504 hours), n=7, 6 | 5.6 (6.16) | 9.5 (7.77)

21. Secondary Outcome: Change From Baseline of Clinical Chemistry Parameters: Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameter including protein at indicated time points. Day -1 value was defined as Baseline for clinical chemistry parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Gram per liter
  24 hours, n=7, 7 | -4.9 (4.06) | -2.3 (4.03)
  96 hours, n=7, 7 | -4.6 (6.80) | -2.9 (1.95)
  168 hours, n=7, 7 | -3.6 (7.32) | -4.1 (2.67)
  336 hours, n=7, 7 | -4.4 (6.29) | -2.4 (1.99)
  Follow-up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow-up (504 hours), n=7, 6 | -5.4 (4.69) | -4.2 (3.54)

22. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet and Leukocytes
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet and leukocytes at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value. Data was not available as all basophil values were below the detection limit. Hence, the change from baseline in basophil values were not calculated.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
10^9 cells per liter
  Basophils, 24 hours, n=0, 0: number analyzed (Participants) | 0 | 0
  Basophils, 96 hours, n=0, 0: number analyzed (Participants) | 0 | 0
  Basophils, 168 hours, n=0, 0: number analyzed (Participants) | 0 | 0
  Basophils, 336 hours, n=0, 0: number analyzed (Participants) | 0 | 0
  Basophils, Follow up (504 hours), n=0, 0: number analyzed (Participants) | 0 | 0
  Eosinophils, 24 hours, n=4, 3: number analyzed (Participants) | 4 | 3
  Eosinophils, 24 hours, n=4, 3 | -0.03 (0.096) | 0.07 (0.058)
  Eosinophils, 96 hours, n=4, 3: number analyzed (Participants) | 4 | 3
  Eosinophils, 96 hours, n=4, 3 | -0.03 (0.150) | 0.00 (0.100)
  Eosinophils, 168 hours, n=4, 3: number analyzed (Participants) | 4 | 3
  Eosinophils, 168 hours, n=4, 3 | 0.00 (0.115) | 0.00 (0.100)
  Eosinophils, 336 hours, n=3, 3: number analyzed (Participants) | 3 | 3
  Eosinophils, 336 hours, n=3, 3 | 0.00 (0.100) | 0.00 (0.100)
  Eosinophils, Follow up (504 hours), n=4, 2: number analyzed (Participants) | 4 | 2
  Eosinophils, Follow up (504 hours), n=4, 2 | -0.05 (0.058) | -0.05 (0.071)
  Lymphocytes, 24 hours, n=7, 7 | -0.27 (0.528) | 0.36 (0.251)
  Lymphocytes, 96 hours, n=7, 7 | -0.11 (0.508) | 0.30 (0.277)
  Lymphocytes, 168 hours, n=7, 7 | -0.10 (0.574) | 0.26 (0.276)
  Lymphocytes, 336 hours, n=7, 7 | -0.50 (0.616) | 0.09 (0.363)
  Lymphocytes, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Lymphocytes, Follow up (504 hours), n=7, 6 | -0.41 (0.441) | 0.00 (0.514)
  Monocytes, 24 hours, n=7, 7 | -0.11 (0.107) | 0.04 (0.113)
  Monocytes, 96 hours, n=7, 7 | -0.04 (0.190) | -0.01 (0.227)
  Monocytes, 168 hours, n=7, 7 | 0.01 (0.186) | 0.00 (0.153)
  Monocytes, 336 hours, n=7, 7 | -0.09 (0.177) | 0.00 (0.115)
  Monocytes, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Monocytes, Follow up (504 hours), n=7, 6 | -0.06 (0.172) | -0.03 (0.216)
  Neutrophils, 24 hours, n=7, 7 | -0.63 (0.939) | -0.54 (0.702)
  Neutrophils, 96 hours, n=7, 7 | -0.76 (1.066) | -0.79 (0.799)
  Neutrophils, 168 hours, n=7, 7 | -0.61 (1.128) | -0.69 (0.546)
  Neutrophils, 336 hours, n=7, 7 | -0.93 (1.181) | -0.96 (0.516)
  Neutrophils, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Neutrophils, Follow up (504 hours), n=7, 6 | -1.09 (1.299) | -0.97 (0.612)
  Platelet, 24 hours, n=7, 7 | -18.3 (18.82) | -11.6 (27.99)
  Platelet, 96 hours, n=7, 7 | -15.1 (20.82) | -6.3 (22.65)
  Platelet, 168 hours, n=7, 7 | -20.0 (26.58) | -13.3 (38.84)
  Platelet, 336 hours, n=7, 7 | -22.4 (35.09) | -27.3 (38.70)
  Platelet, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Platelet, Follow up (504 hours), n=7, 6 | -22.9 (31.49) | -24.3 (44.96)
  Leukocytes, 24 hours, n=7, 7 | -1.00 (1.441) | -0.09 (0.912)
  Leukocytes, 96 hours, n=7, 7 | -0.89 (1.624) | -0.46 (1.149)
  Leukocytes, 168 hours, n=7, 7 | -0.67 (1.738) | -0.36 (0.735)
  Leukocytes, 336 hours, n=7, 7 | -1.50 (1.649) | -0.77 (0.911)
  Leukocytes, Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Leukocytes, Follow up (504 hours), n=7, 6 | -1.59 (1.757) | -0.97 (1.159)

23. Secondary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes
Description: Blood samples were collected for the analysis of hematology parameter including reticulocytes at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Proportion of reticulocytes in blood
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Proportion of reticulocytes in blood
  24 hours, n= 7, 7 | -0.0016 (0.00172) | 0.0003 (0.00125)
  96 hours, n=7, 7 | 0.0017 (0.00544) | -0.0006 (0.00162)
  168 hours, n=7, 7 | 0.0013 (0.00577) | 0.0009 (0.00212)
  336 hours, n= 7, 7 | -0.0011 (0.00430) | 0.0003 (0.00335)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | -0.0013 (0.00368) | 0.0017 (0.00308)

24. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter including hematocrit at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Proportion of red blood cells in blood
  24 hours, n= 7, 7 | 0.001 (0.0135) | 0.007 (0.0198)
  96 hours, n=7, 7 | 0.009 (0.0186) | -0.006 (0.0127)
  168 hours, n=7, 7 | -0.004 (0.0181) | -0.006 (0.0162)
  336 hours, n= 7, 7 | -0.014 (0.0190) | -0.016 (0.0215)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | -0.036 (0.0230) | -0.025 (0.0152)

25. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including hemoglobin at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Gram per liter
  24 hours, n= 7, 7 | 2.0 (2.45) | 3.0 (5.23)
  96 hours, n=7, 7 | 2.6 (5.71) | 0.0 (2.24)
  168 hours, n=7, 7 | 0.0 (5.32) | -1.7 (5.50)
  336 hours, n= 7, 7 | -4.9 (4.95) | -3.6 (4.54)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | -12.1 (6.47) | -6.0 (3.22)

26. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including mean corpuscular hemoglobin at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Picogram
  24 hours, n= 7, 7 | 0.0 (0.00) | 0.0 (0.00)
  96 hours, n=7, 7 | -0.4 (0.53) | 0.0 (0.58)
  168 hours, n=7, 7 | 0.0 (0.82) | -0.1 (0.69)
  336 hours, n= 7, 7 | 0.1 (0.90) | -0.3 (0.76)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | 0.0 (0.58) | -0.2 (0.41)

27. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of hematology parameter including mean corpuscular volume at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Femtoliter
  24 hours, n= 7, 7 | -0.6 (0.98) | -0.7 (2.43)
  96 hours, n=7, 7 | 0.1 (0.90) | -1.4 (1.40)
  168 hours, n=7, 7 | -0.3 (1.11) | -1.1 (1.35)
  336 hours, n= 7, 7 | 0.4 (0.98) | -1.9 (1.68)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | 0.4 (1.27) | -1.7 (1.21)

28. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameter including erythrocytes at indicated time points. Day -1 value was defined as Baseline for hematology parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Day -1), 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
10^12 cells per liter
  24 hours, n= 7, 7 | 0.026 (0.0820) | 0.100 (0.1943)
  96 hours, n=7, 7 | 0.101 (0.1642) | 0.006 (0.0680)
  168 hours, n=7, 7 | -0.024 (0.2204) | -0.021 (0.1906)
  336 hours, n= 7, 7 | -0.187 (0.2051) | -0.079 (0.1901)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | -0.411 (0.2032) | -0.183 (0.1229)

29. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameter
Description: The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of can be read as Trace, + and ++ indicating proportional concentrations in the urine sample. Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Day -1, 24, 96, 168, 336 and follow up (504 hours)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Participants
  Ketones, 336 hours, ++ | 2 | 0
  Ketones, 336 hours, trace | 0 | 1
  Ketones, follow up (504 hours), + | 1 | 0
  Occult blood, 336 hours, + | 1 | 0
  Occult blood, follow up, trace | 0 | 1
  Protein, Day -1, trace | 0 | 1
  Protein, 24 hours, trace | 2 | 3
  Protein, 96 hours, trace | 2 | 4
  Protein, 168 hours, trace | 2 | 1
  Protein, 336 hours, trace | 3 | 3

30. Secondary Outcome: Specific Gravity at Indicated Time Points
Description: Urine samples were collected for analysis of specific gravity of urine. Urinary specific gravity is a measure of the concentration of solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine.
Time Frame: Day -1, 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Ratio
  Day -1, n=7, 7 | 1.0127 (0.00856) | 1.0177 (0.00720)
  24 hours, n=7, 7 | 1.0214 (0.00621) | 1.0256 (0.00665)
  96 hours, n=7, 7 | 1.0211 (0.00832) | 1.0236 (0.00550)
  168 hours, n=7, 7 | 1.0211 (0.00821) | 1.0207 (0.00562)
  336 hours, n=7, 7 | 1.0193 (0.00871) | 1.0246 (0.00945)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | 1.0183 (0.00720) | 1.0222 (0.00728)

31. Secondary Outcome: Urine Potential of Hydrogen (pH) at Indicated Time Points
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Day -1, 24, 96, 168, 336 hours and follow up (504 hours)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
pH
  Day -1, n=7, 7 | 6.21 (0.699) | 6.86 (1.144)
  24 hours, n=7, 7 | 5.86 (0.244) | 5.79 (0.567)
  96 hours, n=7, 7 | 5.79 (0.393) | 6.07 (0.345)
  168 hours, n=7, 7 | 5.93 (0.535) | 6.07 (0.450)
  336 hours, n=7, 7 | 6.00 (0.577) | 6.00 (0.408)
  Follow up (504 hours), n=7, 6: number analyzed (Participants) | 7 | 6
  Follow up (504 hours), n=7, 6 | 6.43 (0.673) | 6.08 (0.492)

32. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), 4, 12, 24, 48, 72, 96, 120, 144, 168, 336 and 504 hours
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Millimeter of mercury (mmHg)
  DBP, 4 hours, n=7, 7 | -7.0 (6.98) | -0.7 (6.92)
  DBP, 12 hours, n=7, 7 | -5.4 (6.02) | -0.3 (8.60)
  DBP, 24 hours, n=7, 7 | -3.9 (5.24) | -2.9 (4.74)
  DBP, 48 hours, n=7, 7 | -3.4 (6.50) | 2.0 (2.08)
  DBP, 72 hours, n=7, 7 | -4.0 (9.11) | -4.6 (5.13)
  DBP, 96 hours, n=7, 7 | -5.9 (10.14) | -2.7 (9.29)
  DBP, 120 hours, n=7, 7 | -4.1 (10.02) | -3.4 (11.16)
  DBP, 144 hours, n=7, 7 | -7.6 (8.81) | -5.4 (7.32)
  DBP, 168 hours, n=7, 7 | -5.1 (10.25) | -1.0 (6.68)
  DBP, 336 hours, n=7, 7 | -5.7 (9.66) | -5.3 (4.39)
  DBP, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  DBP, 504 hours, n=7, 6 | -7.3 (8.73) | -0.7 (10.01)
  SBP, 4 hours, n=7, 7 | -0.1 (5.93) | 1.3 (7.04)
  SBP, 12 hours, n=7, 7 | 1.4 (3.41) | 1.0 (9.73)
  SBP, 24 hours, n=7, 7 | -1.0 (6.32) | -3.4 (11.03)
  SBP, 48 hours, n=7, 7 | -1.9 (6.20) | -1.1 (8.55)
  SBP, 72 hours, n=7, 7 | -1.0 (6.78) | -4.6 (11.80)
  SBP, 96 hours, n=7, 7 | -1.4 (9.96) | 2.6 (8.48)
  SBP, 120 hours, n=7, 7 | -6.3 (5.53) | 0.9 (7.88)
  SBP,144 hours, n=7, 7 | -6.6 (7.30) | -3.3 (6.52)
  SBP, 168 hours, n=7, 7 | 0.4 (8.18) | 0.9 (6.67)
  SBP, 336 hours, n=7, 7 | -3.9 (11.05) | -2.6 (8.81)
  SBP, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  SBP, 504 hours, n=7, 6 | -5.0 (7.92) | -1.5 (5.89)

33. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), 4, 12, 24, 48, 72, 96, 120, 144, 168, 336 and 504 hours
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Beats per minute
  4 hours, n=7, 7 | 3.6 (5.19) | 4.7 (6.95)
  12 hours, n=7, 7 | 5.0 (11.45) | 10.1 (6.74)
  24 hours, n=7, 7 | 3.4 (8.38) | -5.0 (4.36)
  48 hours, n=7, 7 | 3.4 (18.12) | -0.3 (4.39)
  72 hours, n=7, 7 | 4.9 (11.26) | -0.3 (4.15)
  96 hours, n=7, 7 | 1.4 (13.44) | 0.6 (3.21)
  120 hours, n=7, 7 | 1.1 (9.58) | 2.0 (6.11)
  144 hours, n=7, 7 | 0.1 (16.74) | -0.1 (3.24)
  168 hours, n=7, 7 | 4.4 (17.62) | 7.1 (7.20)
  336 hours, n=7, 7 | 1.0 (17.61) | 1.6 (7.50)
  504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  504 hours, n=7, 6 | -2.1 (18.52) | 2.2 (6.79)

34. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), 4, 12, 24, 48, 72, 96, 120, 144, 168, 336 and 504 hours
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Celsius
  4 hours, n=7, 7 | -0.01 (0.195) | 0.27 (0.095)
  12 hours, n=7, 7 | 0.04 (0.172) | 0.26 (0.230)
  24 hours, n=7, 7 | -0.07 (0.150) | -0.01 (0.241)
  48 hours, n=7, 7 | -0.16 (0.190) | -0.04 (0.113)
  72 hours, n=7, 7 | -0.10 (0.271) | -0.10 (0.100)
  96 hours, n=7, 7 | -0.11 (0.212) | -0.04 (0.098)
  120 hours, n=7, 7 | -0.10 (0.191) | -0.17 (0.189)
  144 hours, n=7, 7 | -0.14 (0.223) | -0.09 (0.107)
  168 hours, n=7, 7 | -0.09 (0.186) | 0.01 (0.135)
  336 hours, n=7, 7 | -0.27 (0.315) | -0.13 (0.170)
  504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  504 hours, n=7, 6 | -0.26 (0.479) | -0.07 (0.242)

35. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval, and QT Interval Corrected for Heart Rate by Fredericia's Formula (QTcF) Interval
Description: A single 12-lead ECG was obtained at indicated time points using an ECG machine that automatically measures PR, QRS, QT, and QTcF intervals. Day 1 (Pre-dose) value was defined as Baseline for ECG parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), 4, 12, 24, 48, and 504 hours
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Millisecond
  PR Interval, 4 hours, n=7, 7 | -5.3 (4.07) | -4.6 (5.44)
  PR Interval, 12 hours, n=7, 7 | -8.7 (10.52) | -5.9 (3.89)
  PR Interval, 24 hours, n=7, 7 | -3.1 (8.67) | -0.1 (5.70)
  PR Interval, 48 hours, n=7, 7 | -17.0 (33.80) | 0.3 (5.41)
  PR Interval, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  PR Interval, 504 hours, n=7, 6 | -7.3 (10.05) | 2.2 (9.91)
  QRS duration, 4 hours, n=7, 7 | -1.6 (1.40) | -2.1 (3.24)
  QRS duration, 12 hours, n=7, 7 | -0.3 (3.86) | -0.6 (4.04)
  QRS duration, 24 hours, n=7, 7 | 0.3 (2.50) | -2.0 (3.96)
  QRS duration, 48 hours, n=7, 7 | 3.1 (11.16) | 0.4 (7.91)
  QRS duration, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  QRS duration, 504 hours, n=7, 6 | -0.3 (3.59) | -0.8 (8.08)
  QT interval, 4 hours, n=7, 7 | -4.0 (15.59) | -20.4 (14.28)
  QT interval, 12 hours, n=7, 7 | -17.9 (29.17) | -21.7 (20.09)
  QT interval, 24 hours, n=7, 7 | 4.3 (25.79) | -7.3 (7.48)
  QT interval, 48 hours, n=7, 7 | 2.3 (21.55) | -14.7 (13.50)
  QT interval, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  QT interval, 504 hours, n=7, 6 | 14.7 (32.07) | -9.2 (22.93)
  QTcF interval, 4 hours, n=7, 7 | -4.9 (10.42) | -6.6 (12.39)
  QTcF interval, 12 hours, n=7, 7 | -7.7 (8.94) | -5.7 (12.72)
  QTcF interval, 24 hours, n=7, 7 | -0.9 (7.71) | -0.1 (12.76)
  QTcF interval, 48 hours, n=7, 7 | 11.6 (40.64) | -2.9 (12.88)
  QTcF interval, 504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  QTcF interval, 504 hours, n=7, 6 | 6.7 (12.84) | -2.2 (9.64)

36. Secondary Outcome: Change From Baseline of ECG Parameter: ECG Mean Heart Rate
Description: A single 12-lead ECG was obtained at indicated time points using an ECG machine that automatically calculates mean ECG heart rate. Day 1 (Pre-dose) value was defined as Baseline for ECG parameters. Change from Baseline was defined as difference between post-dose visit values minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), 4, 12, 24, 48, and 504 hours
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
Number analyzed (Participants) | 7 | 7
Beats per minute
  4 hours, n=7, 7 | -2.3 (11.37) | 6.0 (6.32)
  12 hours, n=7, 7 | 2.3 (19.91) | 7.1 (5.37)
  24 hours, n=7, 7 | -5.3 (19.67) | 3.1 (6.72)
  48 hours, n=7, 7 | 6.7 (15.64) | 5.0 (5.32)
  504 hours, n=7, 6: number analyzed (Participants) | 7 | 6
  504 hours, n=7, 6 | -7.1 (25.71) | 3.2 (7.65)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected up to Day 23
Description: Non-serious AEs and SAEs for Safety Population was reported
Arm/Group | Healthy Japanese Participants | Healthy Caucasian Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Japanese Participants (N=7) | Healthy Caucasian Participants (N=7)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03258762/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03258762/SAP_001.pdf